CLINICAL TRIAL: NCT04816656
Title: An Integrated Digital PROM-platform for Cancer Patients During the COVID-19 Pandemic
Acronym: COVID-ONCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Collaborators: Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20.60-onco20.07
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Oncology; PROMs; Chemotherapeutic Toxicity
Keywords: Digital Health; Telemonitoring; Supportive Cancer Care; Oncology; PROMs; COVID-19
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): All patients were presented the digital PROMs platform during their chemotherapy
  Interventions: Other: ePROMs assessment

INTERVENTIONS:
Other: ePROMs assessment — At inclusion the patient received a unique login code which he/she used to start the care path. After signing the informed consent on the digital pathway, the patient needed to fill in the questionnaires that were presented at fixed time points throughout this study.
  Based on the data collected from the questionnaires the patient received customized information and advice. In case of COVID-19, the information and advice was based on the guidelines from Sciensano and the Belgian government. If the patient suffered from side effects from the cancer therapy, they received tips and tricks how to manage these complications. The collected data was forwarded to the patient medical file. As such health care workers were be able to use this information in the patients' follow up consultations.
  Other Names: Digital PROMs platform

SUMMARY:
During the COVID-19 pandemic, patients with cancer are subject to multiple risks (e.g. frequent hospital visits, increased infection risk, more severe clinical course, discontinued cancer treatment etc.).

Patients undergoing cancer therapy are also faced with several Quality of Life - impairing side effects. In the case of a positive COVID-19 cancer patient, the need and intensity of treating must be weighed against the possible higher risk of developing severe complications in the course of a COVID-19 infection. Nevertheless, both for COVID-19 positive and negative patients who will continue or discontinue cancer treatment throughout the pandemic, providing supportive care is more important than ever.

Digitally monitoring patient-reported outcome measures (PROMs) could offer a solution to improve the supportive care measures during cancer treatment, and certainly in times of COVID-19. Digitalized PROMS could significantly contribute to improved communication, patient satisfaction, supportive care, monitoring of cancer treatment, and detection of problems.

To date, clinical trials investigating the benefits of digital PROMS in patients with cancer during the current COVID-19 pandemic are lacking.

At the Jessa Hospital, the investigators already have experience in collecting PROMs via a digital platform (Awell Health) since 2019 for patients with breast cancer undergoing chemotherapy using validated QoL questionnaires.

The overall aim of this project is to prospectively evaluate the impact of a COVID-19 infection on the severity of the cancer therapy-related complications and the QoL of patients with cancer undergoing chemotherapy using a digital PROMs-platform.

DETAILED DESCRIPTION:
General aim: The overall aim of this project is to prospectively evaluate the impact of a COVID-19 infection on the severity of the cancer therapy-related complications and the QoL of patients with cancer undergoing chemotherapy using a digital PROMs platform.

Objective 1: Evaluate the effect of a COVID-19 infection on the severity of cancer therapy-related side effects and patients' QoL

Rationale: The functionality of this platform will be based on three main principles:

1. The digital PROMs platform will provide patient-tailored information throughout the course of their disease and up to one month after the end of their chemotherapy concerning complications and COVID-19. This will support the cancer patients during their disease with specific advice based on the side effects they document. First, this will help comfort patients and reduce their anxiety and insecurity in these stressful times. Second, they will receive information regarding measures they can take to tackle their specific complications. Third, this will encourage patients to seek help in case of a possible COVID-19 infection and/or severe side effects by contacting the oncological support team or their physician.
2. The platform will prospectively collect QoL data using validated patient-reported questionnaires and specific COVID-19 questionnaires via a mobile application.
3. The platform will be fully integrated into the electronic health record (EHR) of the patient and will provide a structured report of the questioned complications for the physician. This will allow the medical oncologist to monitor the medical journey of the patient during and up to one month after their chemotherapy. As such, the medical oncologist can finetune the cancer treatment and supportive care measures towards the needs of the patient.

Hypothesis: "An COVID-19 infection will aggravate the severity of the cancer therapy-related complications and thereby diminish the patients' QoL."

Objective 2: Evaluate the patient benefit of digital PROMS platform Rationale: The implementation of a digital PROMs platform for cancer patients has demonstrated multiple benefits in the past, ranging from enhanced patient satisfaction, detection of unrecognized problems, earlier detection of complications, and/or more specific supportive care measures leading to an improved treatment outcome and QoL.

Hypothesis: "The use of a digital PROMs platform for cancer patients undergoing chemotherapy during the COVID-19 pandemic will lead to (1) an improved patient satisfaction and general knowledge on the oncologic supportive care measures and (2) a reduction in patient distress and anxiety".

General approach (for both objectives): A prospective, cohort study will be set up in patients with cancer undergoing chemotherapy. Patients will be stratified during treatment in two groups: (1) COVID-19 positive and (2) negative patients. Patients will be instructed to fill in validated Qol, distress/anxiety, and COVID-19 specific questionnaires via a digital platform from the day of inclusion up to 1-month post-chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with any type of cancer (except breast cancer)
* Undergoing or starting chemotherapy with or without surgery
* Age ≥ 18 years
* Access to the online application via computer or smartphone
* Able to comply with the study protocol
* Able to sign written informed consent in the digital AWELL platform
* Provide a signed informed consent

Exclusion Criteria:

* Diagnosed with breast cancer and undergoing chemotherapy (patients are already included in the healthcare path breast at Jessa Hospital)
* Undergoing other therapies (e.g. immunotherapy, radiotherapy, targeted therapy, hormonal therapy)
* Insufficient understanding of the Dutch language
* Severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Baseline
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 1 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 2 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 3 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 4 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 5 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 6 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 7 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 8 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 9 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 10 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 11 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 12 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 13 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 14 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 15 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 16 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 17 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 18 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 19 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 20 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 21 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 22 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 23 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Week 24 of chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | 1 week post-chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | 2 weeks post-chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | 3 weeks post-chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | 1 month post-chemotherapy
  Questionnaire to evaluate the presence and severity of therapy-related side effects
5-level EQ-5D version (EQ5D5L) | Baseline
  Questionnaire to evaluate patients' health-related quality of life on five different levels
5-level EQ-5D version (EQ5D5L) | Month 1 of chemotherapy
  Questionnaire to evaluate patients' health-related quality of life on five different levels
5-level EQ-5D version (EQ5D5L) | Month 2 of chemotherapy
  Questionnaire to evaluate patients' health-related quality of life on five different levels
5-level EQ-5D version (EQ5D5L) | Month 3 of chemotherapy
  Questionnaire to evaluate patients' health-related quality of life on five different levels
5-level EQ-5D version (EQ5D5L) | Month 4 of chemotherapy
  Questionnaire to evaluate patients' health-related quality of life on five different levels
5-level EQ-5D version (EQ5D5L) | Month 5 of chemotherapy
  Questionnaire to evaluate patients' health-related quality of life on five different levels
5-level EQ-5D version (EQ5D5L) | Month 6 of chemotherapy
  Questionnaire to evaluate patients' health-related quality of life on five different levels
5-level EQ-5D version (EQ5D5L) | 1 month post-chemotherapy
  Questionnaire to evaluate patients' health-related quality of life on five different levels
Covid-19 triage questionnaire | Baseline
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 1 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 2 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 3 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 4 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 5 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 6 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 7 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 8 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 9 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 10 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 11 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 12 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 13 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 14 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 15 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 16 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 17 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 18 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 19 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 20 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 21 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 22 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 23 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | Week 24 of chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | 1 week post-chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | 2 weeks post-chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | 3 weeks post-chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
Covid-19 triage questionnaire | 1 month post-chemotherapy
  Questionnaire to screen patients for the possibility of a COVID-19 infection.
COVID-19 questionnaire | First day of positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Second day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Third day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Fourth day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Fifth day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Sixth day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Seventh day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Eight day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Ninth day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Tenth day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Eleventh day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Twelfth day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Thirteenth day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 questionnaire | Fourteenth day after positive COVID-19 test
  Questionnaire about symptom burden related to COVID-19
COVID-19 Peritraumatic Distress Index (CPDI) | Baseline
  Questionnaire to capture the frequency of specific phobias and stress disorders relevant to COVID-19, including anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behavior, physical symptoms and loss of social functioning
COVID-19 Peritraumatic Distress Index (CPDI) | Month 1 of chemotherapy
  Questionnaire to capture the frequency of specific phobias and stress disorders relevant to COVID-19, including anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behavior, physical symptoms and loss of social functioning
COVID-19 Peritraumatic Distress Index (CPDI) | Month 2 of chemotherapy
  Questionnaire to capture the frequency of specific phobias and stress disorders relevant to COVID-19, including anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behavior, physical symptoms and loss of social functioning
COVID-19 Peritraumatic Distress Index (CPDI) | Month 3 of chemotherapy
  Questionnaire to capture the frequency of specific phobias and stress disorders relevant to COVID-19, including anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behavior, physical symptoms and loss of social functioning
COVID-19 Peritraumatic Distress Index (CPDI) | Month 4 of chemotherapy
  Questionnaire to capture the frequency of specific phobias and stress disorders relevant to COVID-19, including anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behavior, physical symptoms and loss of social functioning
COVID-19 Peritraumatic Distress Index (CPDI) | Month 5 of chemotherapy
  Questionnaire to capture the frequency of specific phobias and stress disorders relevant to COVID-19, including anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behavior, physical symptoms and loss of social functioning
COVID-19 Peritraumatic Distress Index (CPDI) | Month 6 of chemotherapy
  Questionnaire to capture the frequency of specific phobias and stress disorders relevant to COVID-19, including anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behavior, physical symptoms and loss of social functioning
COVID-19 Peritraumatic Distress Index (CPDI) | 1 month post-chemotherapy
  Questionnaire to capture the frequency of specific phobias and stress disorders relevant to COVID-19, including anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behavior, physical symptoms and loss of social functioning
Patient satisfaction | Month 1 of chemotherapy
  Questionnaire to evaluate their general satisfaction and the user friendliness of the digital platform and how it improved their supportive care
Patient satisfaction | Month 2 of chemotherapy
  Questionnaire to evaluate their general satisfaction and the user friendliness of the digital platform and how it improved their supportive care
Patient satisfaction | Month 3 of chemotherapy
  Questionnaire to evaluate their general satisfaction and the user friendliness of the digital platform and how it improved their supportive care
Patient satisfaction | Month 4 of chemotherapy
  Questionnaire to evaluate their general satisfaction and the user friendliness of the digital platform and how it improved their supportive care
Patient satisfaction | Month 5 of chemotherapy
  Questionnaire to evaluate their general satisfaction and the user friendliness of the digital platform and how it improved their supportive care
Patient satisfaction | Month 6 of chemotherapy
  Questionnaire to evaluate their general satisfaction and the user friendliness of the digital platform and how it improved their supportive care
Patient satisfaction | 1 month post-chemotherapy
  Questionnaire to evaluate their general satisfaction and the user friendliness of the digital platform and how it improved their supportive care

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, MD, PhD, Principal Investigator — Jessa Hospital
Locations (2):
- Belgium (2):
  - Hasselt University, Hasselt, Limburg
  - Jessa Ziekenhuis, Hasselt, Limburg